CLINICAL TRIAL: NCT02329912
Title: The SmartPill® as an Objective Parameter to Evaluate Severity and Duration of Postoperative Ileus
Brief Title: Postoperative Ileus: Duration and Severity Assessment With the SmartPill®
Acronym: PIDuSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Collaborators: University of Bonn (Other)
Responsible Party: Principal Investigator, Dr. med. Tim Vilz, Deputy Head of the Surgical Study Center, University Hospital, Bonn
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHI-201202; O-112.0055 (Other Grant/Funding Number: BONFOR)
Record Dates: First submitted 2014-12-01; First posted 2015-01-01 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Postoperative Ileus
Keywords: postoperative ileus; SmartPill; gastrointestinal transit; prokinetic drugs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients after abdominal surgery (Experimental): SmartPill application after abdominal surgery
  Interventions: Device: SmartPill
- Patients after extraabdominal surgery (Sham Comparator): SmartPill after extraabdominal surgery
  Interventions: Device: SmartPill

INTERVENTIONS:
Device: SmartPill — Application of the SmartPill at the end of surgery

SUMMARY:
Postoperative ileus (POI) is a frequent complication after abdominal surgery leading to nausea, vomiting and infectious complications. Bowel dysmotility can last for days and necessitates parenteral nutrition resulting in an prolonged hospital stay and a high economic burden.

Until now there is no evidence based therapy of manifest POI because of missing valid surrogate markers demonstrating the severity and resolution of POI.

A novel tool to examine gastrointestinal function is the SmartPill®. By measuring pH value, temperature and intraluminal pressure the capsule is able to analyse gastric emptying, small bowel transit, large bowel transit and peristaltic activity.

Unfortunately the use of the SmartPill® is not allowed in the first three months after abdominal surgery. Therefore a trial is needed to investigate the behaviour of the SmartPill® during its passage through the human gastrointestinal tract immediately after surgery.

The primary endpoint is

- to investigate the safety of the SmartPill® in patients after abdominal surgery.

The secondary endpoints are:

* is the SmartPill® able to detect the gastrointestinal transit and the peristaltic activity followed by abdominal surgery compared with patients which underwent thoracic/vascular surgery.
* is it possible to correlate the measured parameters (delayed gastrointestinal transit, lack of peristalsis) with the clinical signs of POI (nausea, vomiting, prolonged duration until first postoperative defecation).
* is the detected peristaltic activity influenced by intravenous applicated prokinetic drugs
* is the detected peristaltic activity influenced by physiotherapy

Using those endpoints the investigators hope to demonstrate the safety of the SmartPill® after abdominal surgery, to evaluate its ability to analyse severity and length of POI and to examine whether the used prokinetic drugs and postoperative mobilization are able to influence peristaltic activity.

DETAILED DESCRIPTION:
Postoperative ileus (POI) is a frequent complication after abdominal surgery leading to nausea, vomiting and infectious complications. Bowel dysmotility can last for days and necessitates parenteral nutrition resulting in an prolonged hospital stay and a high economic burden.

Until now there is no evidence based therapy of manifest POI. Instead, the quality of the existing clinical trials are just of low or moderate quality. The main reason for this is the lack of a valid surrogate marker to define the end of POI: Some trials used first flatus or first defecation as a marker for purposeful peristalsis and resolution of POI, others used the ability to consume solid food again or auscultation of bowel sounds. However it remains questionable whether these parameters are really able to demonstrate the severity or the end of POI.

Therefore POI research needs a reliable, patient and investigator independent parameter that is able to determine resolution of POI to improve the quality of future clinical trials.

A novel tool to examine gastrointestinal function is the SmartPill®. The capsule is able to measure pH value, temperature and intraluminal pressure after oral application, the data is sent to a transmitter located near the patient. Using those values, it is possible to analyse gastric emptying, length of small bowel, large bowel or whole gut passage and the smooth muscle contractility/peristalsis of the whole gastrointestinal tract. Therefore the SmartPill® would be an ideal, patient and investigator independent tool to investigate gastrointestinal function and transit time after visceral surgery.

Unfortunately the use of the SmartPill® is not allowed in the first three months after abdominal surgery. Therefore a trial is needed to investigate the behaviour of the SmartPill® during its passage through the human gastrointestinal tract immediately after surgery.

The primary endpoint is

- to investigate the safety of the SmartPill® in patients after abdominal surgery.

The secondary endpoints are:

* is the SmartPill® able to detect the gastrointestinal transit and the peristaltic activity followed by abdominal surgery compared with patients which underwent thoracic/vascular surgery.
* is it possible to correlate the measured parameters (delayed gastrointestinal transit, lack of peristalsis) with the clinical signs of POI (nausea, vomiting, prolonged duration until first postoperative defecation).
* is the detected peristaltic activity influenced by intravenous applicated prokinetic drugs
* is the detected peristaltic activity influenced by physiotherapy

Using those endpoints the investigators hope to demonstrate the safety of the SmartPill® after abdominal surgery, to evaluate its ability to analyse severity and lenght of POI and to examine whether the used prokinetic drugs and postoperative mobilization are able to influence peristaltic activity.

ELIGIBILITY:
Inclusion Criteria:

* abdominal surgery or thoracic/periphery vascular surgery with an estimated operation time > 90 min and < 10 h
* Age > 18 years
* written informed consent
* ASA score I - III
* negative serum pregnancy test

Exclusion Criteria:

* allergy against the device or components of the device
* existing or planned pregnancy
* emergency surgery
* NSAID (non steroidal antiinflammatory drugs) induced enteropathy
* BMI > 40
* dysphagia
* medical history of gastric bezoars
* medication with proton pump inhibitor, H2-blockers or antacids
* necessity of an MRI in the first two weeks after the operation
* ASA score IV or higher
* gastro-esophageal reflux ("Savary and Miller" III or IV)
* anastomosis between esophagus and jejunum
* fistula or stenosis of the GI tract which is not treated by the operation
* active Crohn´s disease
* Diverticulitis/severe diverticulosis, which is not treated during the operation
* the following operations: all kind of organ transplantations, extended liver resections (extended right or left hemihepatectomy), very low rectum resection with or without a loop ileostoma, small bowel resection with end-to-end anastomosis, near total gastrectomy, transhiatal extended gastrectomy
* patients undergoing abdominal surgery with an increased bleeding propensity (INR > 2, thrombocytes < 50 G/l...)
* perioperative treatment with ciclosporin, tacrolimus, sirolimus, everolimus, methotrexate, Decortin > 15 mg/d, bevazicumab
* no complete inspection for adhesions, fistulas etc. was possible during the operation
* unexpected events during the operation (major bleeding with transfusion of 2 or more erythrocyte concentrates, hazardously anastomosis) mentioned by the surgeon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-03 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
ADEs / SADEs in Patients after surgery | Participants will be followed from first postoperative day until excretion of the SmartPill, an expected average of 8 days
  Number of participants with ADEs / SADEs in Patients after surgery

SECONDARY OUTCOMES:
Analysis of pH value measured by the SmartPill during gastrointestinal passage | Participants will be followed from first postoperative day until excretion of the SmartPill, an expected average of 8 days
  Analysis of pH changes measured by the SmartPill during gastrointestinal passage
Correlation between clinical signs of POI resolution and passage time of the SmartPill | Participants will be followed from first postoperative day until excretion of the SmartPill, an expected average of 8 days
  Analysis of the correlation between clinical signs of targeted peristalsis (time until first defecation in combination with tolerance of solid food) and gastric emptying (hours), small bowel and large bowel transit time (hours)
Peristaltic activity before and after application of prokinetics | Participants will be followed from first postoperative day until excretion of the SmartPill, an expected average of 8 days
  Variation of intraluminal pressure and peristaltic waves (mmHg) measured by the SmartPill before and after intravenous application of prokinetic drugs
Peristaltic activity before, during and after physiotherapy | Participants will be followed from first postoperative day until excretion of the SmartPill, an expected average of 8 days
  Variation of intraluminal pressure and peristaltic waves (mmHg) measured by the SmartPill before, during, and one hour after physiotherapy
Analysis of pressure measured by the SmartPill during gastrointestinal passage | Participants will be followed from first postoperative day until excretion of the SmartPill, an expected average of 8 days
  Analysis of pressure changes (mmHg) measured by the SmartPill during gastrointestinal passage
Analysis of temperature measured by the SmartPill during gastrointestinal passage | Participants will be followed from first postoperative day until excretion of the SmartPill, an expected average of 8 days
  Analysis of temperature changes (°C) measured by the SmartPill during gastrointestinal passage

CONTACTS AND LOCATIONS:
Overall Officials: Tim O. Vilz, MD, Study Director — Department of Surgery, University of Bonn
Locations (1):
- Department of Surgery, University of Bonn, Bonn, Germany

REFERENCES:
- [Background] Tran K, Brun R, Kuo B. Evaluation of regional and whole gut motility using the wireless motility capsule: relevance in clinical practice. Therap Adv Gastroenterol. 2012 Jul;5(4):249-60. doi: 10.1177/1756283X12437874. PMID 22778790
- [Background] Storch I, Barkin JS. Contraindications to capsule endoscopy: do any still exist? Gastrointest Endosc Clin N Am. 2006 Apr;16(2):329-36. doi: 10.1016/j.giec.2006.01.017. PMID 16644461
- [Derived] Vilz TO, Pantelis D, Lingohr P, Fimmers R, Esmann A, Randau T, Kalff JC, Coenen M, Wehner S. SmartPill(R) as an objective parameter for determination of severity and duration of postoperative ileus: study protocol of a prospective, two-arm, open-label trial (the PIDuSA study). BMJ Open. 2016 Jul 8;6(7):e011014. doi: 10.1136/bmjopen-2015-011014. PMID 27401360